CLINICAL TRIAL: NCT02334839
Title: The Association Between Severity of Hypertensive Disorder During Pregnancy and Endothelial Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Liran hiersch, MD, Rabin Medical Center
Other Study IDs: 0206-14
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Endothelial Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Preeclampsia: women with diagnosed preeclampsia
  Interventions: Other: Observational only
- gestational hypertension: women with diagnosed gestational hypertension without preeclampsia
  Interventions: Other: Observational only
- healthy: women without gestational hypertension or preeclampsia
  Interventions: Other: Observational only

INTERVENTIONS:
Other: Observational only — Endothelial function will be assessed using ENDO-PAT (Itamar medical LTD, Caesarea, Israel) device, which evaluates the change in peripheral vascular tone in reaction to temporal ischemia in a process called Reactive Hyperemia (RH) .The RH-PAT is a blood pressure measurement-like cuff which is placed on the non-dominant arm. A pneumatic probe is placed on the index finger bilaterally (one serves as a control). After a baseline assessment for a 5 minutes period, the cuff is inflated to a 60mm Hg pressure above the systolic pressure in order to occlude the arterial flow distal to the brachial artery. After 5 minutes of occlusion, a prompt deflation of the cuff results in a RH response and vasodilatation in the distal arteries including those monitored in the index finger. The sensor translates the change in vascular tone and the ENDO-PAT V3.0.4 device analyzes the data automatically. The results are given in a RH index scale that reflects the level of reactive hyperemia.

SUMMARY:
Preeclampsia toxemia (PET) is a pregnancy related complication that is usually expressed as new onset hypertension and proteinuria after 20 weeks of gestation. scarce data exists regarding the effectiveness of PAT plethysmography use in women with PET and whether adverse results are found compared to healthy gravidas. Thus, we aimed to assess endothelial function using PAT plethysmography in women with PET and compare their results to both healthy gravidas and those with only gestational hypertension.

.

DETAILED DESCRIPTION:
Preeclampsia toxemia (PET) is a pregnancy related complication that is usually expressed as new onset hypertension and proteinuria after 20 weeks of gestation. Although the exact pathophysiology is unclear, it's related to abnormal placentation and subsequent vascular pathology. Endothelial dysfunction was found to play a significant role in the risk of cardiovascular event in general. Moreover, few studies found a relation between endothelial dysfunction and PET. There are several methods for the assessment of endothelial function, with Peripheral Artery Tone (PAT) plethysmography being an emerging non-invasive promising technique. However, scarce data exists regarding the effectiveness of PAT plethysmography use in women with PET and whether adverse results are found compared to healthy gravidas.

Thus, we aimed to assess endothelial function using PAT plethysmography in women with PET and compare their results to both healthy gravidas and those with only gestational hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age 18-40 years old
2. 27 and above weeks of gestation
3. Singleton pregnancy
4. Agreed to participate in the study and signed on informed consent form.

Exclusion Criteria:

1. Known ischemic heart disease or angina pectoris
2. Active smoker
3. Dyslipidemia, chronic hypertension. Renal disease, diabetes mellitus (gestational or pregestational)
4. Active treatment with anti-hypertensive medication, anti-aggregation medication or lipid lowering agents.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A prospective cohort study of approximately 150 gravidas who are hospitalized in maternal-fetal medicine (MFM) ward in Rabin Medical Center in Israel.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Reactive Hyperemia Index (RHI) | 24 months
  The difference in Reactive Hyperemia Index (RHI) as messureas using the ENDOPAT device between the study groups

CONTACTS AND LOCATIONS:
Overall Officials: Liran Hiersch, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin medical center, Petah Tikva, Israel